CLINICAL TRIAL: NCT00761670
Title: Comparative Efficacy of Amisulpride vs Risperidone on Cognitive Functions in Patients With Chronic Schizophrenia
Brief Title: Efficacy Study on Cognitive Functions in Schizophrenic Patients
Acronym: AMIMIND
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMISU_L_01008; EudraCT #: 2007-005772-13
Record Dates: First submitted 2008-09-26; First posted 2008-09-29 (Estimated); Last update posted 2010-12-09 (Estimated); Status verified 2010-12

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Amisulpride; Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: amisulpride and risperidone
- 2 (Active Comparator)
  Interventions: Drug: amisulpride and risperidone

INTERVENTIONS:
Drug: amisulpride and risperidone — amisulpride tablet 400-800 mg/day risperidone tablet 4-8 mg/day

SUMMARY:
Primary objectives

* To compare neurocognitive effects of amisulpride with those of risperidone in patients with chronic schizophrenia, as assessed by the general cognitive index, a measure of overall cognitive functioning in schizophrenia

Secondary objectives

* Secondary analyses will be conducted to determine how the two atypical agents' neurocognitive effects compare with regard to their profile of therapeutic action (based on individual cognitive domain scores in seven cognitive domains, including speed of processing, attention/vigilance, working memory, verbal learning and memory, visual learning and memory, reasoning and problem solving and social cognition);
* Investigate whether amisulpride elicits more improvement on negative symptoms compared to risperidone treatment, as measured by the total score on the Scale of the Assessment of Negative Symptoms (SANS) 8 and by the Negative Symptom Subscale of the Positive and Negative Symptom Scale (PANSS);
* Assess whether amisulpride improves overall functioning and individual domains of psychotic symptoms compared to risperidone as measured by the Clinical Global Impression (CGI), and the total and positive and general psychopathology subscale scores of PANSS and by the individual domains of SANS, respectively;
* Evaluate the safety and tolerability of amisulpride and risperidone based on the study completion rates, and frequency of abnormal laboratory values, prolactin serum concentrations and on the Simpson Angus Scale for Extrapyramidal Symptoms (SAS) 10 and the Abnormal Involuntary Movement Scale (AIMS).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: DSM-IV schizophrenia (any subtype)
* Duration of illness: ≥ 5 years
* Concomitant standing or prn medications (except other antipsychotics and those contraindicated in the respective package inserts [amisulpride or risperidone]) are permitted during treatment phase, if they were present at a stable dose for at least 6 weeks prior to the start of initial treatment with study medication
* Overall symptom severity: patients must evidence a total score of 60 or higher on the PANSS scale
* Clinical Symptoms: A score of 4 (moderate) or greater on any of the 7 items of the PANSS Positive Symptom Subscale is present
* Cognitive status (minimum performance level): subject must be able to validly complete the baseline MATRICS assessment
* Clinical judgment by the investigator that treatments with amisulpride or risperidone are warranted due to suboptimal clinical outcome despite previous treatments

Exclusion Criteria:

* Past or current intolerance of amisulpride or risperidone side effects that are judged by the investigator to be unsafe, dose-limiting, or likely to result in study discontinuation.
* Any contraindication for amisulpride or risperidone therapy as indicated in the drug description.
* Presence of any unstable or untreated medical disorder.
* Any history of seizures or seizure disorder other than febrile seizures of childhood;
* History of positive hepatitis B surface antigen.
* Any abnormal laboratory test that is judged to be clinically significant by the investigator.
* A history of significant head injury/trauma, as defined by:

A. loss of consciousness (LOC) for more than 1 hour B. recurring seizures resulting from the head injury C. clear cognitive sequelae of the injury D. cognitive rehabilitation following the injury

* Alcohol or substance dependence within the past 12 months or abuse within the past 3 months. Any subject with positive urine toxicology or alcohol use that is considered abnormal at baseline.
* Clinically significant suicidal or homicidal behavior or attempts within past 6 months.
* Pregnant or breast-feeding women
* Absence of medically approved contraceptive methods for female of childbearing potential.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2008-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
General cognitive index, as assessed by the overall average z-score based on the neurocognitive test (MATRICS) battery | Day 0, Day 28, Day 56

SECONDARY OUTCOMES:
Cognitive measures assessed by individual subscales scores in seven cognitive domains | Day 0, Day 28, Day 56
Overall Clinical Effects assessed by the Clinical Global Impression (CGI) | Day -21 to -1, Day 0, Day 7, Day 28, Day 56
Clinical symptoms Ratings of psychopathology assessed by the PANSS (positive and negative symptoms, general psychopathology), and the SANS (Attention, Affect, Alogia, asociality/Anhedonia;Avolition) | Day -21 to -1, Day 0, Day 7, Day 28, Day 56
Ratings of potential side affects assessed by the Simpson-Angus Scale (SAS)and the Abnormal Involuntary Movement Scale (AIMS) | Day 0, Day 7, Day 28, Day 56
General safety/tolerability assessed by vital signs measures, treatment emergent adverse events record, and frequency of abnormal laboratory measures | Day -21 to -1, Day 0, Day 28, Day 56

CONTACTS AND LOCATIONS:
Overall Officials: László Erős, MD, Study Director — sanofi-aventis Hungary
Locations (1):
- Sanofi-Aventis Administrative Office, Budapest, Hungary